CLINICAL TRIAL: NCT04404777
Title: Local Recurrence Due to Rectal Cancer in Sweden - the Actual Incidence, Treatment and Outcome After Treatment
Brief Title: Local Recurrence Due to Rectal Cancer in Sweden
Acronym: LERIS
Status: Active, not recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, PI, Sahlgrenska University Hospital
Other Study IDs: LERIS
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Therapeutics; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with local recurrence
  Interventions: Procedure: Treatment for local recurrence with surgery or other treatments

INTERVENTIONS:
Procedure: Treatment for local recurrence with surgery or other treatments — All types of treatment for local recurrence will be evaluated

SUMMARY:
The aim of this retrospective national registry study is to validate the reporting of local recurrence in the registry. Another aim is to identify preoperative risk factors for local recurrence. This can in turn indicate the need for a more intense follow-up. The treatment of local recurrence, including the impact of the multidisciplinary team conference (MDT) and the surgical procedure and the referral pathways of local recurrences will also be determined.

We aim to evaluate treatment outcome after local recurrence for patients operated or treated between 2007-2018.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer with a curative intent

Exclusion Criteria:

* Rectal cancer without curative intent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients treated in Sweden with a curative intent in 2007-2018 will be included. The number of recurrences, patterns of recurrence and outcome after treatment will be evaluated
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of local recurrences | Between 2007-2018
3 year survival | 3 years

SECONDARY OUTCOMES:
Percentage R0 resection after local recurrence | 1-2 months after initiated treatment
MDT effect on treatment of local recurrence | 1-3 months after diagnosis of recurrence
Reported metastases | 5 years
  Number of patients with metastasis reported vs actual
MRI features at primary diagnosis and relation to recurrence | 2 months
  MRI evaluation by radiologist related to recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided